CLINICAL TRIAL: NCT06291155
Title: Molecular Mechanisms of SGLT2 Inhibition in Diabetic Kidney Disease
Brief Title: Mechanism of SGLT2 Inhibition in the Kidney
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Colorado, Denver (Other); Renal Pre-Competitive Consortium (RPC3) (Unknown)
Responsible Party: Principal Investigator, Markus Bitzer, Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00222335
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes; Diabetic Kidney Disease
Keywords: Kidney biopsy; Kidney MRI; SGLT2 inhibitor; SGLT2i; FDA-approved; Renal biopsy; Renal MRI; Type 2 diabetes; Canagliflozin; INVOKANA
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — Sodium-Glucose Transporter 2 Inhibitors; Canagliflozin

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized mechanistic trial of an FDA-approved drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SGLT2i Arm (Other)
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — All participants will be receive 100 mg/daily doses of Canagliflozin (INVOKANA) for 6 months. Canagliflozin is a Sodium-glucose cotransporter 2 (SGLT2) inhibitor
  Other Names: Canagliflozin; Invokana

SUMMARY:
The goal of this open-label, non-randomized clinical trial is to determine what effects, if any, an FDA-approved drug class known as SGLT2 inhibitors (Canagliflozin or INVOKANA) has any protective effects on kidney function in Type 2 diabetes. We are looking for participants 18-80 years of age, who have had a clinical diagnosis of Type 2 diabetes for ≥ 3 years.

Participants will be asked to sign a consent and complete a screening visit prior to study entry including the following procedures for this study:

Consent and Screening:

* Laboratory tests to determine baseline health
* Ultrasound to measure kidney size and ensure presence of 2 functioning kidneys

Month 0:

* Study entry kidney MRI (day 0)
* Study entry kidney biopsy (within 30 days of MRI)
* Study entry visit for dispensing 100 mg/daily Canagliflozin medication 3 month supply

Month 3:

* Study visit to dispense remaining 3 months of 100 mg/daily Canagliflozin medication
* Review of systems

Month 6:

* Follow-up kidney MRI
* Follow-up kidney biopsy

Study participants will also be requested to provide blood and urine samples for biobanking purposes. They will also be provided the opportunity to provide a stool sample at two time points, as well as the option to participate in a related study collecting samples to create induced Pluripotent Stem Cells (iPSCs).

Participants will be compensated for their time and loss of work time, additionally, a nominal additional compensation for optional stool and iPSC samples.

DETAILED DESCRIPTION:
The purpose of this protocol is to examine the effects of the sodium-glucose cotransporter 2 (SGLT2) inhibitor canagliflozin on intrarenal transcripts of energy metabolism in adults with type 2 diabetes and early diabetic kidney disease (DKD) via an open-label non-randomized mechanistic trial. This trial will enroll 40 participants who will receive 100 mg of canagliflozin daily for six (6) months in addition to standard of care. The primary objective of this study is to determine whether canagliflozin affects intrarenal transcripts of energy metabolism in adults with type 2 diabetes and early DKD.

The primary outcomes measure will be change in transcripts as assessed by single-cell RNA sequencing of kidney biopsy specimens obtained at study entry and after 6 months of study drug. Secondary outcomes include assessing the effects of canagliflozin on structural progression of DKD assessed by morphometric examination of kidney tissue specimens from the paired research biopsies. Additional secondary outcomes include measures of glomerular filtration rate (GFR) and renal plasma flow (RPF) as well as multiparametric kidney MRI. Magnetic resonance imaging of the kidneys will be performed prior to each biopsy to correlate the molecular and structural damage seen at kidney biopsy with the level of perfusion, oxygen availability and fibrosis detected by imaging. Imaging of the kidneys will be done as near to the time of each kidney biopsy as possible. Participants will be followed annually after completion of the mechanistic clinical trial until death or development of end-stage kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years.

  * The lower age limit was set so renal function test results would not reflect changes associated with growth.
* Diagnosis of type 2 diabetes for ≥ 3 years.
* Estimated GFR >45 and < 90 ml/min/1.73m2 as determined from the CKD-EPI equation using serum creatinine (Levey et al., 2009)
* A screening urinary albumin-to-creatinine ratio <3000 mg/g.
* Willingness to participate after receiving a thorough explanation of the study.
* Participants receiving a RAAS inhibitor must have been receiving the drug at maximum tolerable dose for at least 3 months prior to the study baseline examination.
* Participants receiving a GLP-1 receptor agonist must have been receiving the drug for at least 3 months prior to the study baseline examination.
* Participants must meet the current clinical guidelines for prescribing SGLT2 inhibitors, to maintain FDA-approved standards

Exclusion Criteria:

* Clinically significant disorders of the liver [cirrhosis, portal hypertension, hepatitis, increased bilirubin (≥1.5 mg/dl), active or uncontrolled cardiovascular disease, symptomatic peripheral vascular disease, (i.e. intermittent claudication), pulmonary diseases (including uncontrolled asthma and restrictive or obstructive lung disease requiring therapy), renal-urinary disorders (calculi, urinary tract obstruction, glomerulonephritis, chronic infection), gastrointestinal disorders (nausea, vomiting, diarrhea or anorexia sufficient to cause weight loss or wasting), or hematocrit levels ≤30 percent in women or ≤35 percent in men.
* Prior and ongoing treatment with SGLT2 inhibitors
* Renovascular or malignant hypertension; uncontrolled hypertension (systolic blood pressure ≥150 or diastolic ≥90 mm Hg)
* Hematuria of unknown etiology.

  * Prior to entry into the study, any participant with hematuria should be evaluated, the etiology established and documented, and treatment rendered as appropriate.
* Chronic debilitating disorders with or without treatment (e.g., systemic lupus erythematosus [SLE], cancer, amyloidosis, and chronic infection) that would interfere with the assessment of kidney function or that might reduce the chances of survival for a sufficient length of time to evaluate the efficacy of treatment.
* Currently receiving a drug regimen that includes steroids, immunosuppressants, or investigational new drugs not associated with this trial.
* Pregnancy.

  * SGLT2 inhibitors are not recommended during the second or third trimester of pregnancy. Moreover, we do not wish to expose pregnant women to conscious sedation that is used during the kidney biopsies.. Women of childbearing potential must have a negative pregnancy test prior to entry and every 2 months during the study and agree to using an effective form of contraception throughout the study, such as the oral contraceptive pill or an intrauterine device. Women who are planning a pregnancy in the next three years will be excluded.
* Known hypersensitivity to canagliflozin or iodine.
* Bleeding disorders or requirements for anticoagulation or platelet inhibitors which cannot be safely interrupted since kidney biopsies cannot be performed safely in these individuals.
* Massive obesity with body mass index ≥45 kg/m².

  * Kidney biopsies are more technically difficult with massive obesity.
* Allergy to iodine-containing contrast material or shellfish.
* Non-diabetic kidney disease - based on clinical history or kidney biopsy examination.
* History of osteoporotic fracture.
* History of lower-limb amputation irrespective of etiology
* Conditions likely to interfere with informed consent or compliance with the protocol.
* Known solitary kidney
* Size of one or both kidneys on ultrasound < 9 cm (small kidney size is concerning for renal atrophy due to underlying kidney disease) or > 2 cm discrepancy between left and right kidney sizes based on largest longitudinal diameter
* Current use of UGT enzyme inducters, lithium, and digoxin
* Blood urea nitrogen (BUN) > 80 gm/dL
* INR > 1.4 (a)
* PTT > 35 seconds (a)
* Platelet count < 100,000 uL (a)
* Hemoglobin (Hgb) < 10 mg/dL (a)
* Hydronephrosis or other important renal ultrasound findings such as significant stone disease

  1. Inclusion possible after this has been obtained within range

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Glomerular basement membrane (GBM) width and mesangial expansion | Baseline and 6 months
  Measured by morphometric examination of kidney tissue

SECONDARY OUTCOMES:
Kidney Transcript Changes | 6 month follow-up
  Molecular changes measured by change in transcripts as assessed by single-cell RNA sequencing of kidney biopsy specimens

CONTACTS AND LOCATIONS:
Overall Officials: Markus Bitzer, MD, Principal Investigator — Professor of Internal Medicine
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No